CLINICAL TRIAL: NCT03217981
Title: Sepse: Critical Analysis of New Sepse Studies and Definitions and Retrospective Evaluation of Sepse Protocol Implementation at Hospital Unimed Volta Redonda
Brief Title: Sepse: Critical Analysis of New Sepse Definitions and Retrospective Evaluation of Sepse Protocol at a Tertiary Hospital in Brazil
Acronym: HUVR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unimed Volta Redonda (Other)
Responsible Party: Principal Investigator, Vicente Lopes da Silva Junior, Principal Investigator, Unimed Volta Redonda
Other Study IDs: HUVR17.1
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2015: 2015 - Individuals with a diagnosis of sepsis from June 2014 to May 2015
  Interventions: Other: Sepsis protocol
- 2016: 2016 -Individuals with a diagnosis of sepsis from June 2015 to May 2016
  Interventions: Other: Sepsis protocol

INTERVENTIONS:
Other: Sepsis protocol — Adherence to the sepsis protocol

SUMMARY:
Research in the databases Lilacs, BIREME, SciELO by the terms: systemic inflammatory response syndrome (SIRS), sepsis, severe sepsis and septic shock and their equivalents in the English language. Selection of the main articles of the last five years to study and contextualize the reality presented since the implantation of the HUVR sepsis protocol. Statistical analysis of data since the implementation of the sepsis protocol in the HUVR, in July 2014 until June 2016.

ELIGIBILITY:
Inclusion Criteria:

All individuals who had a confirmed or suspected sepsis diagnosis and had a sepsis protocol completed during the study period.

-

Exclusion Criteria:

Individuals with confirmed or suspected sepsis in the study period who did not complete the protocol.

Individuals under the age of 18

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age hospitalized with suspected or confirmed diagnosis of sepsis at HUVR.
Sampling Method: Non-Probability Sample
Enrollment: 506 (Estimated)
Dates: Start 2017-08-02 (Actual); Primary Completion 2017-08-05 (Estimated); Study Completion 2017-08-08 (Estimated)

PRIMARY OUTCOMES:
Adherence to the sepsis protocol | From 2014 to 2016
  Implementation of the measures recommended in the sepsis protocol

SECONDARY OUTCOMES:
Sepsis mortality rate | From 2014 to 2016
  Assessment of the evolution of the sepsis mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Leila Auler, Study Director — Director
Locations (1):
- Vicente Lopes, Volta Redonda, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No